CLINICAL TRIAL: NCT03451500
Title: Carbidopa-Levodopa in Dry Age Related Macular Degeneration With Geographic Atrophy
Brief Title: Carbidopa-Levodopa in Dry AMD With Geographic Atrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding required for enrollment to reach statistical significance.
Sponsor: Snyder, Robert W., M.D., Ph.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0004
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Age Related Macular Degeneration
Keywords: GPR 143; PEDF; VEGF; LDOPA
MeSH Terms: conditions — Macular Degeneration | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, placebo controlled
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All tablets will be identical in appearance. The Director of Research will be aware of treatment assignment. Patients, their Care Providers and all other study staff will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Carbidopa-levodopa 2 tablets daily (Experimental): carbidopa-levodopa 25-100 mg 2 tablets daily hs
  Interventions: Drug: carbidopa-levodopa
- carbidopa-levodopa 6 tablets daily (Experimental): carbidopa-levodopa 25-100 mg, 2 tablets, 3 times daily, with breakfast, with supper and hs
  Interventions: Drug: carbidopa-levodopa
- Placebo (Placebo Comparator): Placebo, 2 tablets, 3 times daily, with breakfast, with supper and hs
  Interventions: Drug: carbidopa-levodopa

INTERVENTIONS:
Drug: carbidopa-levodopa — See previous

SUMMARY:
From 3 large patient databases, patients diagnosed with AMD who have never taken levodopa(L-DOPA) containing medications have a mean age of diagnosis at 71 years.

Patients who have been treated with L-DOPA containing medications have a mean age of diagnosis of AMD at 79 years. L-DOPA binds to GPR143 in the retinal pigment epithelium, and releases PEDF, which protects the retina and downregulates VEGF, which is the cause of neovascularization.

The Investigators will evaluate the safety and tolerability of carbidopa-levodopa in patients with Neovascular AMD, and measure the effects on visual acuity and retinal abnormalities due to "wet" (neovascular) AMD. The Investigators will evaluate the safety and tolerability of carbidopa-levodopa in patients with Dry AMD and Geographic Atrophy, and measure the effects on visual acuity, area of geographic atrophy and other retinal abnormalities due to "dry" AMD.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the most common cause of blindness, in individuals over the age of 50, in the developed world. AMD becomes more common as people age, and is more common in lightly pigmented individuals. AMD appears more common in patients with Parkinson's Disease, than in those without. The AREDS nutritional supplements are effective in slowing the progress of intermediate AMD(5).

Most AMD is "dry AMD", which progresses relatively slowly and may impair vision, but usually does not lead to legal blindness. There are two forms of AMD, "wet AMD" and geographic atrophy (GA), that can cause more profound vision loss. In aggregate they occur in about 25% patients with AMD. Wet AMD is due to new growth of abnormal blood vessels under the retina. The new blood vessels are believed to be due to an excessive release of vascular endothelial growth factor (VEGF) by the retinal pigment epithelium(RPE) cells. Wet AMD is now effectively treated with intraocular injections of VEGF inhibitors. Geographic Atrophy, the other form of advanced AMD, represents focal death of the RPE cells and overlying neurosensory retina. There is no current treatment for GA. It is suspected that GA is due in part to a localized inflammatory response, damage to RPE cells and loss of RPE cell function. It may also be speculated that stimulation of RPE cells to release a potent neurotrophic factor, pigment epithelium derived factor (PEDF) may slow progression of GA. In 2008, Dr. Brian McKay identified a receptor, G protein coupled receptor

#143(GPR143), on the surface of RPE cells and discovered that L-DOPA was the natural ligand or stimulator of GPR143. Dr McKay showed that treatment of RPE cells with exogenous L-DOPA resulted in the release of additional PEDF. In subsequent work Dr McKay's group also showed that L-DOPA stimulation of PEDF in RPE cells was also associated with a decrease in VEGF. Thus, Dr McKay hypothesized that exogenous LDOPA may prevent the onset of AMD or progression to wet AMD.

In 2015, Dr McKay and his associates published a paper that showed that patients, who had been treated with L-DOPA, had a delay in the onset of AMD by 8 years, compared to patients who had not been treated with L-DOPA. In addition, those who had AMD and went on to develop wet AMD, did so 5 years later than those with no history of L-DOPA treatment. L-DOPA is an intermediate in the pigmentation pathway. Dr McKay and his associates suggested that the reason darkly pigmented races do not get AMD nearly as frequently as lighter pigmented races, is that they produce more pigment, and thus more L-DOPA to stimulate GPR143 on RPE cells. According to this hypothesis, the stimulated RPE cells release PEDF and decrease VEGF, which together are responsible for the protective effect.

Pharmacology of L-DOPA and carbidopa:

L-DOPA is formed by 3-hydroxylation of tyrosine by tyrosine-3-monooxygenase (tyrosinase).(18) The primary metabolic pathway of L-DOPA is decarboxylation by amino acid decarboxylase to dopamine, which is responsible for most, but not all, of its pharmacologic effects and toxicity. When carbidopa is administered with LDOPA, systemic levels of L-DOPA double and central nervous system (CNS) L-DOPA increases from about 1% of the administered dose to about 4%. Levodopa freely passes from the systemic circulation into the retina and brain, but dopamine and carbidopa do not. Adverse events are markedly decreased when carbidopa is administered with L-DOPA, because systemic levels of the toxic metabolite of L-DOPA, dopamine, are markedly reduced. In most patients, 25 mg of carbidopa is sufficient to control side effects of 100 mg of L-DOPA, primarily nausea, by 90%. L-DOPA is the natural ligand for GPR143 in the RPE cells. The Investigators' intent is to increase the L-DOPA available to RPE surface receptors (GPR 143) while minimizing peripheral toxicity. This concept is unique, because all other uses of L-DOPA rely on CNS conversion of L-DOPA to dopamine, in order to produce the desired effect.

Since there are no established animal models for AMD, and L-DOPA has a good safety profile in healthy volunteers and patients with Parkinson's disease, the Investigators propose a prospective experiment to determine the safety and tolerability of L-DOPA, in a population of patients with AMD. The participants will be made aware of potential side effects of L-DOPA, which are listed in the Informed Consent, during the consent process. Adverse events will be elicited by questioning the participants at each visit.

The participants will also be advised to call the site, if they have any medical problem between visits.

The Investigators will also use this study to examine whether L-DOPA has a positive effect on visual acuity and pathologic retinal changes of "dry" AMD with geographic atrophy.

The parameters to be evaluated are best corrected ETDRS visual acuity, area of geographic atrophy by Fundus AutoFluorescence (FAF), macular thickness by spectral domain optical coherence tomography (SD OCT), new blood (hemorrhage) by direct retinal examination, and subjective decrease in vision.

Treatments:

Study participants will receive randomly assigned, single blind, commercially available carbidopa-levodopa 25-100 mg, two tablets once daily hs, or two tablets dosed TID (three times daily), in the morning, with supper and hs for one month, or placebo two tablets dosed three times daily, in the morning, with supper and hs (200-600 mg of levodopa daily). This is the equivalent of low to moderate doses of carbidopa-levodopa in patients with Parkinson's disease (daily dose of levodopa 200-800 mg). If a study participant experiences non-serious, but bothersome adverse effects while taking the study medication, the dose may be reduced to 1 tablet hs, or 1 tablet TID.

Number of subjects: 154 randomized.

Duration: 12 months of treatment, with visits at Baseline, 1 week, 1 month, 3 months, 6 months, 9 months and 12 months.

Primary Endpoint: A statistically significant difference in progression of area of geographic atrophy with carbidopa-levodopa treatment compared to treatment with placebo.

Measurements and Activities:

1. Informed Consent at Baseline;
2. Ophthalmic history and comprehensive eye examination; including visual acuity, with best optical correction, using an EDTRS chart, in both eyes prior to randomization, ophthalmoscopic examination, a subjective vision questionnaire and SD OCT with FAF;
3. Repeat assessment of visual acuity using an EDTRS chart, subjective vision questionnaire, ophthalmoscopic examination, and SD OCT at 1, 3, 6 9, and 12 month visits;
4. Demographics at Baseline;
5. Medical History, Vital Signs and Physical Examination at Baseline;
6. ECG, CBC, Chem 20 and HbA1C at Baseline;
7. Dispense study medication at visits 2, 3, 4, 5, 6 and 7;
8. Pill count at visits 3, 4, 5, 6 and 7;
9. Non-directed assessment of adverse events at each visit, including classification as to severity, seriousness and body system.
10. Concomitant medications at each visit.

Statistics: Statistics will be generated for, at a minimum, , area of geographic atrophty, ETDRS visual acuity, central retinal thickness and presence of hemorrhage. Within patient trajectories for these outcomes will be plotted, incorporating information on dose and duration. Analysis of Variance may be conducted to relate logarithm of dose and duration of treatment to the outcomes listed above.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of dry AMD with geographic atrophy in one or both eyes. In patients with geographic atrophy in both eyes, the eye with the larger area of geographic atrophy will be designated eye A and the eye with the smaller area of geographic atrophy will be designated eye B.
2. Normal or dry AMD of any grade in the second eye;
3. Age 50-85 years;
4. Willingness to maintain AREDS vitamin supplements throughout the study, or remain off these supplements for the duration of the study, if not taking them prior to the study;
5. Signed Informed Consent.

Exclusion criteria:

1. Any previous or current use of L-DOPA containing medication or dopamine agonist medication, or any planned use of any of these agents, except for study medication, during the study;
2. Concurrent use of monoamine oxidase (MAO) inhibitors;
3. Any eye condition, disease, or history of trauma in either eye, which can impair vision, except cataract or cataract surgery;
4. BCVA worse than 20/100 in the eye with better BCVA;
5. Current, or history of, neovascular AMD in either eye;
6. Neurologic conditions which can impair vision;
7. Parkinson's Disease;
8. Significant orthostatic hypotension, defined as a drop in systolic blood pressure, immediately upon changing from the supine to standing position, of >19 mmHg, or a symptomatic drop in systolic blood pressure, immediately upon changing from the supine to standing position;
9. Significant ECG abnormalities, as judged by the Investigator;
10. Estimated glomerular filtration rate (eGFR) <20 ml/min;
11. Liver enzymes >3 X the upper limit of normal;
12. HbA1C >9.0;
13. Any other significant lab abnormalities, as judged by the Investigator.
14. Women of childbearing potential;
15. Known retinal hemorrhage;
16. Subjects who are not fluent in English.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Area of Geographic Atrophy | Change over 12 months
  area of retinal geographic atrophy measured by fundus autofluorescence

SECONDARY OUTCOMES:
Best Corrected Visual Acuity by ETDRS | Change over 12 months
  Best Corrected Visual Acuity by ETDRS
Central retinal thickness | Change over 12 months
  Central Retinal Thickness, measured by SD-OCT
Development of neovascular macular degeneration | New diagnosis during 12 months of treatment
  New diagnosis of neovascular macular degeneration

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C Fagan, MD, Study Director — Robert Snyder, MD, PhD, PC; Robert W Snyder, MD, PhD, Principal Investigator — Robert Snyder, MD, PhD, PC
Locations (1):
- Robert W Snyder, MD, PhD, PC, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No